CLINICAL TRIAL: NCT04432077
Title: Piloting an Integrated Anxiety Intervention for Preschool Children With Autism Spectrum Disorder
Brief Title: Anxiety Intervention for Preschool Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Organization for Autism Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019A06
Record Dates: First submitted 2020-06-03; First posted 2020-06-16 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Anxiety Disorder; Autism Spectrum Disorder
MeSH Terms: conditions — Anxiety Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All participants receive the DINOSAUR intervention
  Interventions: Behavioral: DINO Strategies for Anxiety and fear of Uncertainty Reduction (DINOSAUR)

INTERVENTIONS:
Behavioral: DINO Strategies for Anxiety and fear of Uncertainty Reduction (DINOSAUR) — DINO Strategies for Anxiety and fear of Uncertainty Reduction (DINOSAUR) - a parent-mediated cognitive-behavioral treatment modified for young children with ASD

SUMMARY:
This study evaluates the feasibility, acceptability, and preliminary efficacy of a treatment program for anxiety in preschool children with autism spectrum disorder.

DETAILED DESCRIPTION:
Anxiety is highly prevalent in individuals with ASD with lifelong impact. In this population, anxiety often emerges when children are very young, yet there are no evidence-based treatments for this age group. Cognitive-behavioral treatment (CBT) successfully reduces anxiety levels in young, typically developing children and older children with ASD. This study pilots the DINO Strategies for Anxiety and fear of Uncertainty Reduction (DINOSAUR) program, which is an integrated treatment program that utilizes CBT modified for young children with ASD. The treatment includes heavy doses of parent training to reduce accommodation of the child's anxiety symptoms and interventions targeting fear of uncertainty, a common fear in children with ASD. The feasibility, acceptability, and preliminary efficacy of this treatment program will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 years 0 months to 6 years 11 months
* NVIQ ≥ 85 based on Mullen Scales of Early Learning or Stanford Binet 5
* Expressive and Receptive Language scores ≥ 85 based on Preschool Language Scale - Fifth Edition or Orals or Written Language Scales, Second Edition
* DSM-5 diagnoses of Separation Anxiety, Social Anxiety, and/or Generalized Anxiety Disorder and/or the distinct diagnosis of Other Social Fear based on the results of the Anxiety Disorders Interview Schedule/ASA

Exclusion Criteria:

* History of psychological trauma
* History of neurologic illness
* Parent substance abuse, bipolar disorder, psychosis
* Parents require support from a medical interpreter
* Child displays severe behavior challenges
* Severe eyesight or hearing impairments that may interfere with the protocols
* Child's behavior prevents their ability to participate in a 1 hour group consisting of various activities (e.g., listening to a story, snacks, playing movement games, completing a craft)

Ages: 48 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in child anxiety diagnostic status on Anxiety Disorders Interview Schedule, Autism Spectrum Disorder Addendum (ADIS-ASA) after 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (baseline to pre-treatment); Before and after 12-week treatment (pre-treatment to post-treatment)
  clinician administered, semi-structured interview assessing anxiety disorders; clinical severity ratings range from 0 to 3 or 0 to 8; higher scores indicate more impairment
Improvement in child anxiety symptoms on Clinical Global Impressions Scale-Improvement following 12-week intervention | Following 12-week intervention (post-treatment)
  used to assess treatment response; scores range from 1 (very much improved) to 7 (very much worse)

SECONDARY OUTCOMES:
Change in child anxiety symptoms on Preschool Anxiety Scale - Revised following 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (baseline to pre-treatment); Before and after 12-week intervention (pre-treatment to post-treatment)
  parent and teacher report scale measuring levels of anxiety in preschool aged children; scores range from 0 to 112; higher scores indicate higher anxiety
Change in child anxiety symptoms on the Screen for Child Anxiety Related Disorders following 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (baseline to pre-treatment); Before and after 12-week intervention (pre-treatment to post-treatment)
  parent and teacher report scale measuring levels of anxiety in children older than 5 years old; scores range from 0 to 114; higher scores indicate higher anxiety
Change in severity of anxiety and other psychiatric symptoms on Child Behavior Checklist following 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (baseline to pre-treatment); Before and after 12-week intervention (pre-treatment to post-treatment)
  an established 99-item parent and teacher report of broad psychopathology; T scores range from 20 to 100; Syndrome scales: T-scores over 65 indicate clinically significant symptoms
Change in child's tolerance of uncertainty on Response to Uncertainty and Low Environmental Stability Scale following 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (baseline to pre-treatment); Before and after 12-week intervention (pre-treatment to post-treatment)
  parent and teacher report scale measuring response to uncertainty and low environmental structure; scores range from 1 to 5; higher scores indicate higher intolerance of uncertainty
Change in child ASD symptoms on Social Responsiveness Scale following 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (baseline to pre-treatment); Before and after 12-week intervention (pre-treatment to post-treatment)
  parent report scale that assesses the presence and severity of social impairment in children; T-scores range from 20 to 100; higher scores indicate higher ASD severity
Change in child repetitive behaviors on Repetitive Behavior Scale-Revised following 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (baseline to pre-treatment); Before and after 12-week intervention (pre-treatment to post-treatment)
  parent-report measure of repetitive behavior in children with ASD; scores range from 0 to 176; higher scores indicate greater impairment
Change in parental anxiety and depression symptoms on Hospital Anxiety and Depression Scale following 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (baseline to pre-treatment); Before and after 12-week intervention (pre-treatment to post-treatment)
  parental screening tool that captures clinical anxiety and depression; scores range from 0 to 21; higher scores indicate higher anxiety and/or depression symptoms
Change in parental tolerance of uncertainty on Intolerance of Uncertainty Scale following 12-week waitlist and 12-week intervention | Before and after 12-week wailist (baseline to pre-treatment); Before and after 12-week intervention
  parental scale that measures responses to uncertainty, ambiguous situations and the future; scores range from 12 to 60; higher scores indicate higher intolerance of uncertainty
Change on parental accommodating behaviors on Family Accommodation Scale following 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (baseline to pre-treatment); Before and after 12-week intervention (pre-treatment to post-treatment)
  assesses parental accommodating behaviors; scores range from 0 to 36; higher scores indicate higher parental accommodation
Change in child attention bias to threat on Behavioral Paradigms following 12-week waitlist and 12-week intervention | Before and after 12-week waitlist (pre-treatment to post-treatment); Before and after 12-week intervention (pre-treatment to post-treatment)
  eye tracking paradigms used to assess attention bias to threat; more frequent saccades to threatening stimuli indicate higher attention bias to threat

CONTACTS AND LOCATIONS:
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keefer A, Kreiser NL, Singh V, Blakeley-Smith A, Duncan A, Johnson C, Klinger L, Meyer A, Reaven J, Vasa RA. Intolerance of Uncertainty Predicts Anxiety Outcomes Following CBT in Youth with ASD. J Autism Dev Disord. 2017 Dec;47(12):3949-3958. doi: 10.1007/s10803-016-2852-z. PMID 27405445
- [Background] Reaven J, Moody EJ, Grofer Klinger L, Keefer A, Duncan A, O'Kelley S, Meyer A, Hepburn S, Blakeley-Smith A. Training clinicians to deliver group CBT to manage anxiety in youth with ASD: Results of a multisite trial. J Consult Clin Psychol. 2018 Mar;86(3):205-217. doi: 10.1037/ccp0000285. PMID 29504790
- [Derived] Keefer A, Vasa RA. DINOSAUR: an integrated cognitive-behavioral treatment for anxiety in young children with ASD. J Neurodev Disord. 2021 Oct 11;13(1):46. doi: 10.1186/s11689-021-09396-9. PMID 34635048